CLINICAL TRIAL: NCT05755048
Title: A Multicenter, Open-label, Randomized Controlled Phase III Clinical Study to Compare the Efficacy and Safety of FS-1502 Versus T-DM1 in Patients With HER2-positive Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: FS-1502 Versus T-DM1 for HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FS-1502-III1-01
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FS-1502 (Experimental): Experimental: FS-1502 Dosage form: lyophilized powder Specification: 30 mg/vial Dose: 2.3 mg/kg, once every 3 weeks, 21 days as a cycle; Method of administration: intravenous drip.
  Interventions: Biological: Investigational drug: Recombinant Anti-HER2 Humanized Monoclonal Antibody - Monomethyl Auristatin F Conjugates for Injection (FS-1502)
- Trastuzumab Emtansine (T-DM1) (Active Comparator): Active Comparator: Trastuzumab Emtansine (T-DM1) Trade name: Kadcyla Dosage form: lyophilized powder Specification: 100 mg/vial Dose: 3.6 mg/kg, once every 3 weeks, 21 days as a cycle; Method of administration: intravenous drip (this drug has been approved for marketing. Please refer to the package insert for details).
  Interventions: Biological: Control drug: Trastuzumab emtansine (Kadcyla, T-DM1)

INTERVENTIONS:
Biological: Investigational drug: Recombinant Anti-HER2 Humanized Monoclonal Antibody - Monomethyl Auristatin F Conjugates for Injection (FS-1502) — Experimental: FS-1502 Dosage form: lyophilized powder Specification: 30 mg/vial Dose: 2.3 mg/kg, once every 3 weeks, 21 days as a cycle; Method of administration: intravenous drip.
  Arms: FS-1502
Biological: Control drug: Trastuzumab emtansine (Kadcyla, T-DM1) — Active Comparator: Trastuzumab Emtansine (T-DM1) Trade name: Kadcyla Dosage form: lyophilized powder Specification: 100 mg/vial Dose: 3.6 mg/kg, once every 3 weeks, 21 days as a cycle; Method of administration: intravenous drip (this drug has been approved for marketing. Please refer to the package insert for details).
  Arms: Trastuzumab Emtansine (T-DM1)

SUMMARY:
This study is designed to compare the anti-tumor activity as well as the safety and efficacy of FS-1502 versus T-DM1 in HER2-positive, unresectable locally advanced or metastatic breast cancer subjects previously treated with trastuzumab and taxane.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, randomized controlled phase III clinical study to compare the efficacy and safety of FS-1502 versus T-DM1 in patients with HER2-positive unresectable locally advanced or metastatic breast cancer. Patients who meet the inclusion and exclusion criteria will be randomized into the test group (FS-1502) or control group (T-DM1) in a 1:1 ratio. Patients in the test group will receive FS-1502 2.3 mg/kg, and those in the control group will receive T-DM1 3.6 mg/kg, by intravenous drip every 3 weeks. Patients will be treated until disease progression (PD), intolerable toxicity, withdrawal of consent, death, or other protocol-specified reasons. According to the Response Evaluation Criteria in Solid Tumours (RECIST 1.1), tumor assessment will be performed every 6 weeks (± 7 days) for the first 12 months and every 12 weeks (± 7 days) after 12 months until PD, withdrawal of consent, or death. Efficacy evaluation will be performed by the investigator and the Independent Review Committee (IRC), respectively.

ELIGIBILITY:
Inclusion Criteria:Subjects are eligible to be included in the study only if they meet all of the following criteria:

1. Male or female age ≥ 18;
2. Histologically or cytologically confirmed HER2-positive unresectable locally advanced or metastatic breast cancer;
3. Prior treatment with trastuzumabs and taxanes in the adjuvant therapy, neoadjuvant therapy, or advanced treatment phases;
4. ≥ 1 and ≤ 3 previous lines of therapy against locally advanced or metastatic diseases, if PD occurring during adjuvant therapy/neoadjuvant therapy and within 12 months after treatment can be taken as one line of therapy;
5. Tissue samples qualified by the central laboratory for HER2 detection are available, and HER2 is confirmed positive by the pathology test in the central laboratory: Immunohistochemistry (IHC) 3+, or IHC2+ and fluorescence in situ hybridization (FISH)+ as the basis for inclusion;
6. ECOG score at 0 or 1;
7. Expected survival ≥ 12 weeks;
8. Adequate organ and bone marrow functions: absolute neutrophil count [ANC] ≥1.0×10^9/L (no use of granulocyte-colony-stimulating factor (G-CSF) within 7 days); hemoglobin (HGB) ≥ 90 g/L (no red blood cell transfusion within 14 days); platelet count (PLT) ≥ 100×10^9/L (no use of platelet-elevating drugs within 7 days, no platelet transfusion within 14 days); total serum bilirubin (TSB) ≤ 1.5 × upper limit of normal (ULN) or ≤ 3.0 × ULN for patients with Gilbert syndrome; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN; for patients with liver metastases, AST and ALT ≤ 5×ULN; creatinine clearance ≥ 50 mL/min (calculated by Cockroft-Gault formula); blood potassium ≥3.5 mmol/L; albumin ≥ 3 g/dL; left ventricular ejection fraction (LVEF) >50%; urine protein ≤1+ or 24h urine protein quantification <1.0 g;
9. At least one non-intracranial evaluable lesion as assessed by RECIST 1.1;
10. Female patients of childbearing potential must agree to take highly effective contraceptive measures or avoid sexual intercourse during and after the study and within at least 3 months after the last dose of FS-1502 and within at least 7 months after the last dose of T-DM1. Male patients must agree to avoid sexual intercourse, or they and/or any female partners of childbearing potential must take a medically acceptable and effective contraceptive measure, such as double barrier methods, condoms, oral or injectable contraceptives, intra-uterine devices during and after the study and within at least 3 months after the last dose of FS-1502 or within at least 4 months after the last dose of T-DM1;
11. Be able to understand and voluntarily sign the written Informed Consent Form (ICF).

Exclusion Criteria:

Patients that meet any of the following conditions shall not be included in this clinical study:

1. Patients who have received chemotherapy, small molecule targeted drug therapy, endocrinotherapy，radiotherapy, etc. within 14 days or 5 half-lives (whichever is shorter) before administration or who have received major surgical treatment and tumor immunotherapy within 4 weeks before administration or who have received large molecule monoclonal antibody drugs for cancer treatment within 21 days before administration.
2. Patients who have participated in other clinical studies within 4 weeks or 5 half-lives of the drug (whichever is shorter) before administration.
3. Patients who have been previously treated with anti-HER2 ADCs for metastatic diseases.
4. Patients with known hypersensitivity or delayed type hypersensitivity to certain ingredients of T-DM1 or similar drugs, or with known contraindications for the use of T-DM1.
5. Patients with pia maters, spinal cords, brainstem and brain parenchymal metastases; such patients are allowed to be enrolled if all of the following conditions are met:

   1. Patients who have received local treatment and the lesions are stable for more than 6 months;
   2. Patients who have no clinical symptoms and don't need glucocorticoid therapy or other dehydration treatment, and have a stable dose of an antiepileptic drug, if applicable.
6. Patients with a large quantity of clinically uncontrolled pleural effusion, pericardial effusion, or ascites (within 2 weeks prior to the first dose).
7. Unresolved toxic reactions from previous anti-tumor therapy (> NCI-CTCAE 5.0 Grade 1); however, alopecia, neurotoxicity or other toxicity that has converted to chronic and returned to NCI-CTCAE 5.0 Grade ≤ 2, and does not affect the safety of the patient as assessed by the Investigator are allowed to be enrolled.
8. History of non-infectious interstitial lung disease (ILD) / pneumonia, current ILD / pneumonia, or imaging suggestive of suspected moderate-severe ILD / pneumonia at screening.
9. Subjects with corneal epithelial lesions (except mild punctate keratopathy), or other ocular diseases that affect the evaluation of ocular toxicity after the investigational product administration, or unwilling to stop wearing corneal contact lenses during the study.
10. Patients on medications that prolong the QTc interval (mainly Classes Ia, Ic, III anti- arrhythmia medications) or with risk factors for prolonging the QTc interval, such as uncorrectable hypokalemia, inherited long QT syndrome; potential medications for prolonging the QTc interval are presented in Appendix 7.
11. Cardiac function and diseases that meet one of the following conditions:

    1. Mean QTc > 450 ms for males and mean QTc > 470 ms for females averaged from 3 results of 12-lead ECG measurements using the QTcF formula of the ECG instrument at the study site during the screening period;
    2. New York Heart Association (NYHA) Functional Classification ≥ Class 2 congestive heart failure;
    3. Clinically significant arrhythmia (Grade ≥ 2);
    4. History of myocardial infarction or severe arteriovenous thrombotic events within 6 months.
12. Pregnant or breastfeeding women.
13. Known hypersensitivity to any excipients of FS-1502.
14. Active infection requiring systemic therapy.
15. Active hepatitis B (positive for HBV surface antigen and detected with HBV DNA > 1000 IU/mL or meeting the diagnostic criteria for active hepatitis B infection at the study site) or hepatitis C (positive for HCV RNA) and human immunodeficiency viral infection (HIV positive).
16. Any other malignancy diagnosed within 5 years prior to the study, except for early malignancies (carcinoma in situ) that have undergone radical treatment, such as adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ.
17. Any other diseases or conditions considered clinically significant by the investigator that could affect protocol compliance or affect the patient's ability to sign the ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Based on Independent Central Review (ICR) in Participants With HER2-Positive, Unresectable locally advanced or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane. | Up to 28 months.
  Progression-free survival (PFS) by ICR was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.

SECONDARY OUTCOMES:
Overall Survival (OS) in Participants With HER2-Positive, Unresectable locally advanced or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane. | Up to 28 months.
  Overall survival (OS) was defined as the time from the date of first dose of study drug to the date of death due to any cause.
Objective Response Rate (ORR) Based on ICR and Investigator Assessment in Participants With HER2-Positive, Unresectable locally advanced or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane. | Up to 28 months.
  Objective Response Rate (ORR) was defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by ICR and investigator assessment based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR is reported.
Disease control rate (DCR) Based on ICR and Investigator Assessment in Participants With HER2-Positive, Unresectable locally advanced or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane. | Up to 28 months.
  DCR confirmed by IRC or investigator evaluation is defined as the proportion of patients with objective remission (CR or PR) or stable disease (SD) confirmed by IRC or investigator.
Clinical benefit rate (CBR) Based on ICR and Investigator Assessment in Participants With HER2-Positive, Unresectable locally advanced or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane. | Up to 28 months.
  CBR confirmed by IRC or investigator evaluation is defined as the proportion of patients with confirmed CR, PR and SD lasting ≥ 24 weeks evaluated by IRC or investigator according to RECIST version 1.1.
Duration of overall response (DOR) Based on ICR and Investigator Assessment in Participants With HER2-Positive, Unresectable locally advanced or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane. | Up to 28 months.
  Duration of Response (DOR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DOR in participants with confirmed CR/PR based on BICR and investigator assessment is reported.
Progression-Free Survival (PFS) Based on Investigator Assessment in Participants With HER2-Positive, Unresectable locally advanced or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane. | Up to 28 months.
  Progression-free survival (PFS) by investigator assessment was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Treatment-emergent adverse events (TEAEs). | Up to 28 months.
  Type and frequency of treatment-emergent adverse events (TEAEs) with toxicity grades evaluated according to the National Cancer Institute-Common Toxicity Criteria Adverse Event (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (56):
- China (56):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Chinese People's Liberation Army General Hospital fifth Medical Center South ward, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality
  - Chinese People's Liberation Army Army Special Medical Center, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The 900th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army, Fuzhou, Fujian
  - The first affiliated hospital of xiamen university, Xiamen, Fujian
  - The first Hospital of lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Shantou University School of Medicine Affiliated Cancer Hospital, Shantou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences,Shenzhen Center, Shenzhen, Guangdong
  - Guangxi Medical Univesity Cancer Hospital, Nanning, Guangxi
  - The First Afeliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - AnYang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Renmin Hospital Of Wuhan University, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Chenzhou No.1 People's Hospital, Chenzhou, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Nanchang People's Hospital, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning cancer hospital & institute, Shenyang, Liaoning
  - The first hospital of china medical university, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong First Medical University and Shandong Academy of Medical Sciences Shandong Cancer Hospital institute, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Neijiang Second People's Hospital, Neijiang, Sichuan
  - TianJin Medical university Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Henan Cancer Hospital, Zhengzhou, ZHenan